CLINICAL TRIAL: NCT04741256
Title: Implementation of a Standardized Tracheostomy Education Discharge Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other (terminated before study began)
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4320
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
Keywords: Caregiver activation; Caregiver knowledge; Caregiver skills; Caregiver confidence; Tracheostomy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracheostomy discharge protocol (Experimental): All head and neck cancer patients regardless of participation in the study will receive the standard of care: A copy of a tracheostomy education booklet and standardized discharge training for patients and their caregivers by nursing staff during their inpatient stay.
  Research personnel will provide protocol training to the inpatient nurses who are to provide training to caregivers.
  Pre-implementation phase: Eligible "patient" participants identified & healthcare utilization recorded. "Nursing staff" participants complete nursing survey to capture volume of tracheostomy-related questions received.
  Protocol-phase: "Caregiver" participants will complete a survey prior to patient tracheostomy, on day of patient discharge, and one week following discharge
  Post-implementation phase: "Nursing staff" participants will complete an additional survey similar to the one in the pre-implementation phase. EMR will be reviewed for implementation fidelity.
  Interventions: Behavioral: Education booklet & standardized discharge training

INTERVENTIONS:
Behavioral: Education booklet & standardized discharge training — Tracheostomy education booklet and tracheostomy teaching performed by nurses during hospitalization as dictated by the booklet.

SUMMARY:
The purpose of this study is to identify and establish a safe and effective tracheostomy teaching protocol for caregivers. Results of this study will help in the development of a discharge protocol that allows for caregiver confidence and activation in tracheostomy care for patients.

DETAILED DESCRIPTION:
This is a 3-phase, prospective controlled cohort study .

The first "pre-implementation" phase will include assessment of healthcare utilization costs of tracheostomy patients currently and nursing perspective on current caregiver tracheostomy knowledge.

The second "protocol" phase will include assessment of the necessity, acceptability, feasibility, fidelity, safety and effectiveness of a standardized pathway and assessment of the caregiver's activation.

The third "post-implementation" phase will involve assessment of post-implementation tracheostomy-related healthcare utilization costs and nursing perspective on caregiver tracheostomy knowledge.

ELIGIBILITY:
Inclusion Criteria:

Patient participants:

* Diagnosis of malignancy of the head and neck requiring reconstruction and temporary tracheostomy
* No previous record of tracheostomy
* Has an identified family caregiver who is willing to participate
* Has the tracheostomy in place for at least 10 days after discharge

Caregiver participants:

* Family member or friend, who is 18 years or older, of an adult patient described above
* Identified by the patient as his/her primary caregiver who is providing daily assistance

Exclusion Criteria:

* Patients who do not have a caregiver
* Caregivers who are illiterate.
* Caregivers with previous tracheostomy experience.
* Patients who are decannulated from tracheostomy prior to discharge.
* Patients discharged to a skilled nursing facility at the time of discharge.
* Patients who are tolerating continuous tracheostomy capping at time of discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient-Caregiver Activation Survey scores | At time of surgery, an average of 15 minutes
  Caregiver activation in managing their family members' tracheostomy after implementation of a standardized discharge program as measured by the Patient-Caregiver Activation Survey. This is a validated survey assessing caregiver consisting of 13 questions designed to determined confidence in taking care of their loved one. Scores range from 4 to 52, with higher score indicates higher degree of caregiver activation
Patient-Caregiver Activation Survey scores | At discharge (an average of 7 days after surgery), an average of 15 minutes
  Caregiver activation in managing their family members' tracheostomy after implementation of a standardized discharge program as measured by the Patient-Caregiver Activation Survey. This is a validated survey assessing caregiver consisting of 13 questions designed to determined confidence in taking care of their loved one. Scores range from 4 to 52, with higher score indicates higher degree of caregiver activation
Patient-Caregiver Activation Survey scores | At first follow-up (1 week after discharge), an average of 15 minutes
  Caregiver activation in managing their family members' tracheostomy after implementation of a standardized discharge program as measured by the Patient-Caregiver Activation Survey. This is a validated survey assessing caregiver consisting of 13 questions designed to determined confidence in taking care of their loved one. Scores range from 4 to 52, with higher score indicates higher degree of caregiver activation

SECONDARY OUTCOMES:
Feasibility Questionnaire scores | At time of surgery, an average of 15 minutes
  The feasibility questionnaire evaluates the necessity, acceptability and feasibility of the of the implementation of a standardized discharge program. Questions are related to readiness and willingness to participate in tracheostomy care. It will assess feasibility in attending tracheostomy teaching sessions by nurses and their baseline comfort in tracheostomy care and their enthusiasm in learning tracheostomy care. Questionnaire consists of 12 questions, with scores ranging from 12 to 60, with higher scores indicating higher feasibility of tracheostomy protocol implementation.
Patient Reported Outcomes Measurement Information System (PROMIS) short form scores | At time of surgery, an average of 15 minutes
  Safety, as measured by the PROMIS scores - 7-item questionnaire that assess self-reported anxiety in the family caregiver. A higher score correlates with a higher level of anxiety. Scores range from 7 to 25, with higher scores indicating a greater severity of anxiety
Patient Reported Outcomes Measurement Information System (PROMIS) short form scores | At discharge (an average of 7 days after surgery), an average of 15 minutes
  Safety, as measured by the PROMIS scores - 7-item questionnaire that assess self-reported anxiety in the family caregiver. A higher score correlates with a higher level of anxiety. A higher score correlates with a higher level of anxiety. Scores range from 7 to 25, with higher scores indicating a greater severity of anxiety
Patient Reported Outcomes Measurement Information System (PROMIS) short form scores | At first follow-up (1 week after discharge), an average of 15 minutes
  Safety, as measured by the PROMIS scores - 7-item questionnaire that assess self-reported anxiety in the family caregiver. A higher score correlates with a higher level of anxiety. A higher score correlates with a higher level of anxiety. Scores range from 7 to 25, with higher scores indicating a greater severity of anxiety
Preparedness Caregiver Scale (PCS) | At discharge (an average of 7 days after surgery), an average of 15 minutes
  PCS scores - Response categories correspond to the level of preparedness. Scale consists of 9 questions, with scores ranging from 0 to 4 with high score indicating the more prepared the caregiver feels for caregiving.
Preparedness Caregiver Scale (PCS) | At first follow-up (1 week after discharge), an average of 15 minutes
  PCS scores - Response categories correspond to the level of preparedness. Scale consists of 9 questions, with scores ranging from 0 to 4 with high score indicating the more prepared the caregiver feels for caregiving.
Tracheostomy Care Competency Assessment | At discharge (an average of 7 days after surgery), an average of 15 minutes
  Effectiveness will be measured with the tracheostomy care competency assessment. This survey will be an individual's subjective assessment of his or her knowledge of tracheostomy care. A 5-point Likert scale will be used from 1 "strongly disagree" to 5 "strongly agree" and assess different aspects of tracheostomy care outlined during their tracheostomy teaching provided by nurses. This assessment includes 12 questions with scores ranging from from 12 to 60 with higher scores indicating higher competency.
  Results form pre-implementation to post-implementation will be compared using a paired t-test or McNemar tes
Tracheostomy Care Competency Assessment | At first follow-up (1 week after discharge), an average of 15 minutes
  Effectiveness will be measured with the tracheostomy care competency assessment. This survey will be an individual's subjective assessment of his or her knowledge of tracheostomy care. A 5-point Likert scale will be used from 1 "strongly disagree" to 5 "strongly agree" and assess different aspects of tracheostomy care outlined during their tracheostomy teaching provided by nurses. This assessment includes 12 questions with scores ranging from from 12 to 60 with higher scores indicating higher competency.
  Results form pre-implementation to post-implementation will be compared using a paired t-test or McNemar tes
Average tracheostomy-related healthcare utilization costs | Pre-implementation (up to 6 months prior to surgery)
  Effectiveness will be measured with the tracheostomy care competency assessment. This survey will be an individual's subjective assessment of his or her knowledge of tracheostomy care. A 5-point Likert scale will be used from 1 "strongly disagree" to 5 "strongly agree" and assess different aspects of tracheostomy care outlined during their tracheostomy teaching provided by nurses. This assessment includes 12 questions with scores ranging from from 12 to 60 with higher scores indicating higher competency.
  Results form pre-implementation to post-implementation will be compared using a paired t-test or McNemar tes
Average tracheostomy-related healthcare utilization costs | Post-implementation, 30 days after discharge
  Average pre and post-implementation tracheostomy-related healthcare utilization costs
Nursing survey | Pre-implementation (up to 6 months prior to surgery)
  Effectiveness will be measured with the Nursing Survey scores. This is an 11 question survey designed to capture the amount of phone calls nurses receive regarding tracheostomy related questions over the last 6 months.
  Results form pre-implementation to post-implementation will be compared using a paired t-test or McNemar tes
Nursing survey | Post-implementation, 30 days after discharge
  Effectiveness will be measured with the Nursing Survey scores. This is an 11 question survey designed to capture the amount of phone calls nurses receive regarding tracheostomy related questions over the last 6 months.
  Results form pre-implementation to post-implementation will be compared using a paired t-test or McNemar tes
Number of emergency department visits, urgent care or outpatient appointments post-discharge | Post-implementation, 30 days after discharge
  Number of emergency department visits, urgent care or outpatient appointments, relating to post-discharge assessment of feasibility and safety of intervention
Average number of tracheostomy-related phone calls per week post-discharge | Post-implementation, 30 days after discharge
  Post-discharge assessment of feasibility, as measured by average number of tracheostomy-related phone calls per week

CONTACTS AND LOCATIONS:
Overall Officials: Rod Rezaee, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Insignia Health provides rights to the Patient-Caregiver survey. As part of the agreement for access to the survey, they request that at the conclusion of the study we share the entire de-identified dataset. These will not be published by them or shared with another party